CLINICAL TRIAL: NCT05021627
Title: A Multicenter Randomized Controlled Study of Cardiac Autonomic Nerve Improvement and Pacemaker Therapy in Patients With Sinus Bradycardia
Brief Title: Cardiac Autonomic Nerve Improvement and Pacemaker Therapy in Patients With Sinus Bradycardia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Shandong University of Traditional Chinese Medicine (Other); The Second People's Hospital of Yuhuan City (Unknown)
Responsible Party: Principal Investigator, Xu Liu, Professor, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chest 18
Record Dates: First submitted 2021-08-15; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Sinus Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac autonomic nerve modification (Experimental)
  Interventions: Procedure: Cardiac autonomic nerve modification
- Pacemaker (Active Comparator)
  Interventions: Procedure: Pacemaker implantation

INTERVENTIONS:
Procedure: Cardiac autonomic nerve modification — Patients with sinus bradycardia undergoing cardiac autonomic ganglion ablation. Specific anatomic ablation of the 4 major left atrial GP and aorta-superior vena cava (Ao-SVC) GP was performed. Briefly, catheter ablation was performed under the guidance of an electroanatomic mapping system (CARTO,BiosenseWebster,DiamondBar,California). After completed the electroanatomic mapping of the left atrium was complete and pulmonary vein (PV) ostia identified, presumed GP clusters were ablated 1 to 2cm outside the PV-left atrium junctions at the following sites: the left superolateral area (leftsuperior GP[LSGP]), the leftinfer oposterior area(left inferior GP[LIGP]), the right superoanterior area (rightanterior GP[RAGP]), the right inferoposterior area(right inferior GP[RIGP]), and the Ao-SVC fat pad (Ao-SVCGP), and in that sequence.
  Arms: Cardiac autonomic nerve modification
Procedure: Pacemaker implantation — Patients with sinus bradycardia received pacemaker implantation. The patient lay flat on the bed, puncture the subclavian vein and insert two guide wires. Cut the skin under the guide wire to make a skin bag, and stop bleeding accurately to avoid continuous bleeding of the skin bag. The pacemaker electrode is inserted into the heart cavity by guiding the guide wire, one is placed in the ventricle and the other in the atrium, and the corresponding parameters of the electrode, such as pacing threshold, impedance, etc., are measured at the same time. If the parameters are good, fix the electrode, connect the electrode with the pacemaker, place the pacemaker in the skin bag, fix the pacemaker and electrode, suture the skin layer by layer, and the operation is completed.
  Arms: Pacemaker

SUMMARY:
This is a multicenter randomized controlled study. By comparing patients with sinus bradycardia undergoing cardiac autonomic ganglion ablation and pacemaker therapy, and long-term follow-up to evaluate its safety and effectiveness after surgery, in order to evaluate the safety and effectiveness of cardiac autonomic ganglion ablation in the treatment of sinus bradycardia.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years old;
2. Symptomatic sinus bradycardia;
3. Not meet the class I indications for pacemaker implantation.

Exclusion Criteria:

1. Structural heart disease, heart surgery history;
2. Drug-induced SB, sinus pause >2.0 s, positive atropine test, corrected sinus node recovery time (cSNRT) >525 ms;
3. Any atrial or ventricular arrhythmia, or a history of ablation procedures to treat atrial tachyarrhythmias;
4. With Significant congenital heart disease, ejection fraction was <40% measured by echocardiography;
5. Allergic to contrast media;
6. Contraindication to anticoagulation medications;
7. Severe pulmonary disease e.g. restrictive pulmonary disease, chronic obstructive disease (COPD);

9. Poor general health; 10.Life expectancy less than 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Symptom score after operation | 48 months
  Each patient subjectively assessed his or her SB-related symptom, including dizziness, fatigue, and palpitation, on a score of 1 to 10 points (mildtosevere). The total SB-related symptom score for each patient was calculated as the sum of all scores for individual symptoms.

SECONDARY OUTCOMES:
Quality of life score | 48 months
  The Medical Outcomes Study Short-Form 36 Health Survey (SF-36) was used to assess quality of life (QoL) at baseline and 12 months after ablation. The self-administration mode was strictly followed for QoL surveys. TheSF-36 assesses 8 specific QoL domains, namely physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problem, and mental health. For each subscale, scores were transformed to a scale ranging from 0 to 100, with lower scores representing a lower QoL.
Psychological quality score | 48 months
  The Zung Self-Rating Depression Scale is a short self administered survey to quantify the depressed status of a patient. There are 20 items on the scale that rate the four common characteristics of depression: the pervasive effect, the physiological equivalents, other disturbances, and psychomotor activities.
  There are ten positively worded and ten negatively worded questions. Each question is scored on a scale of 1-4 (a little of the time, some of the time, good part of the time, most of the time).